CLINICAL TRIAL: NCT04757012
Title: Pilot Study to Evaluate the Benefits of Preterm Newborn Exposition to a Maternal Voice and Heardbeat Recording During Hospital Stay
Brief Title: Efficacy Study of a Device Allowing Broadcasting Maternal Voice and Heartbeat in Preterm Newborn (CALIPREM)
Acronym: CALIPREM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: En cours; 2020-A01369-30 (Other: ID-RCB Number)
Record Dates: First submitted 2021-01-24; First posted 2021-02-16 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Preterm Newborn
Keywords: Preterm newborn; Maternal voice reccording; NIPE

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calinage exposition (Experimental): exposition to a maternal voice and heartbeat recording during hospital stay for preterm newborns at D2, D4 and D6
  Interventions: Device: calinange
- no exposition (No Intervention): No exposition to a maternal voice and heartbeat recording during hospital stay for preterm newborns at D1, D3 and D5

INTERVENTIONS:
Device: calinange — calinange
  Arms: Calinage exposition

SUMMARY:
The purpose of this study is to evaluate the benefits of an exposition to a maternal voice and heartbeat recording during hospital stay for preterm newborns. For that, we use of a specific neonatal device "Calinange" able to record maternal voice and heartbeats and to restore it with a sound level control. We hypothesize an improvement of the well being of the newborn under Calinange exposition.

DETAILED DESCRIPTION:
Immediately after birth, preterm newborns are immersed in a hostile environment of intensive care unit with light, sound and painful stimulations. Previously, exposure to maternal voice has demonstrated improvement on infants' statements: reduction of bradycardia, desaturation events, improvement of tolerance feeding and sleep. Unfortunatly in most of the N ICU in France, the mothers' presence attendance time is reduced because of the absence of accommodation structure. The use of a specific neonatal device able to daily record maternal voice and hearbeats and to restore it when mother is gone could improve the environment and promote the well-being of the newborn.

ELIGIBILITY:
Inclusion Criteria:

* hospitalised premature newborn in Port-Royal NICU
* age between 3 and 6 daysof life
* gestational age between 27+0 and 31+6 weeks
* hospitalisation in one bed room
* parental consents
* beneficiaries social security scheme

Exclusion Criteria

* occurrence of one or more non-inclusion criteria
* Non-inclusion Criteria:
* Chromosomal abnormality, severe congenital malformation
* Toxic substance consumption during pregnancy
* Sedative medication in progress, High frequencies ventilation in progress
* Neurological damage: intraventricular haemorrhage stage 3 and 4, bilateral and expanse periventricular leukomalacia lesions
* Severe infectious state requiring haemodynamic support (inotropic drugs or hemissucinate)
* Participation to a other intervention research

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability / NIPE Index | Change of the NIPE index before and after intervention. Each baby is his own control. Nipe index is recorded 10 minutes before and 10 minutes after the intervention (Calinange (day 2/4/6) or nothing (day 1/3/5))
  Recorded heart rate

SECONDARY OUTCOMES:
Number of desaturation events | Change of the NIPE index before and after intervention. Each baby is his own control. Nipe index is recorded 10 minutes before and 10 minutes after the intervention (Calinange (day 2/4/6) or nothing (day 1/3/5))
  Change in desaturation events before and after intervention
Number of apnoeic events | Change of the NIPE index before and after intervention. Each baby is his own control. Nipe index is recorded 10 minutes before and 10 minutes after the intervention (Calinange (day 2/4/6) or nothing (day 1/3/5))
  Change in apneic events before and after intervention
Number of bradycardia events | Change of the NIPE index before and after intervention. Each baby is his own control. Nipe index is recorded 10 minutes before and 10 minutes after the intervention (Calinange (day 2/4/6) or nothing (day 1/3/5))
  Change in bradycardia events before and after intervention
Evaluate the benefits for the nurses | To be completed after each use of calinange ether on day 2, 4 and 6
  Evaluation questionnaire
Evaluate the benefits for the mother | At day 7, after the end of intervention
  Satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Juliana PATKAI, MD, Principal Investigator — Service de Médecine et Réanimation néonatales de Port-Royal APHP.Centre - Université de Paris. Site Cochin.
Locations (1):
- NICU of Port-Royal, Maternity of Port-Royal, Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandre C, De Jonckheere J, Rakza T, Mur S, Carette D, Logier R, Jeanne M, Storme L. [Impact of cocooning and maternal voice on the autonomic nervous system activity in the premature newborn infant]. Arch Pediatr. 2013 Sep;20(9):963-8. doi: 10.1016/j.arcped.2013.06.006. Epub 2013 Jul 23. French. PMID 23890732
- [Background] Filippa M, Devouche E, Arioni C, Imberty M, Gratier M. Live maternal speech and singing have beneficial effects on hospitalized preterm infants. Acta Paediatr. 2013 Oct;102(10):1017-20. doi: 10.1111/apa.12356. Epub 2013 Aug 8. PMID 23848529
- [Background] Williamson S, McGrath JM. What Are the Effects of the Maternal Voice on Preterm Infants in the NICU? Adv Neonatal Care. 2019 Aug;19(4):294-310. doi: 10.1097/ANC.0000000000000578. PMID 31335378
- [Background] Provenzi L, Broso S, Montirosso R. Do mothers sound good? A systematic review of the effects of maternal voice exposure on preterm infants' development. Neurosci Biobehav Rev. 2018 May;88:42-50. doi: 10.1016/j.neubiorev.2018.03.009. Epub 2018 Mar 10. PMID 29535067